CLINICAL TRIAL: NCT02951221
Title: A Phase 1, Open-label Study to Evaluate the Relative Bioavailability of Two Formulations of BIIB074 and to Assess the Effect of Food on BIIB074 Pharmacokinetics in Healthy Subjects
Brief Title: New Formulation and Food Effect Study of BIIB074
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 802HV107
Record Dates: First submitted 2016-10-24; First posted 2016-11-01 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Trigeminal Neuralgia (TN); Other Neuropathic Pain
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Treatment sub groups A and B
  Interventions: Drug: BIIB074 Treatment A; Drug: BIIB074 Treatment B
- Cohort 2 (Experimental): Treatment sub groups C and D
  Interventions: Drug: BIIB074 Treatment C; Drug: BIIB074 Treatment D

INTERVENTIONS:
Drug: BIIB074 Treatment A — Lower dose RCF fasted
  Arms: Cohort 1
Drug: BIIB074 Treatment B — Lower dose DCF fasted
  Arms: Cohort 1
Drug: BIIB074 Treatment C — Higher dose DCF fasted
  Arms: Cohort 2
Drug: BIIB074 Treatment D — Higher dose DCF fed
  Arms: Cohort 2

SUMMARY:
The primary objectives of the study are to assess the relative bioavailability of the BIIB074 direct compression formulation (DCF) to the BIIB074 roller compaction formulation (RCF) and to determine the effect of a high-fat meal on the pharmacokinetics (PK) of the BIIB074 DCF. The secondary objective of the study is to assess the safety and tolerability of BIIB074 administered as the DCF following single oral dose administration in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body mass index between 18 and 30 kg/m2, inclusive.
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.
* Ability to consume and tolerate the entire high-fat breakfast within a 30-minute timeframe.

Key Exclusion Criteria:

* History of, or positive test result at Screening for, human immunodeficiency virus (HIV).
* Positive test result at Screening for hepatitis C virus antibody.
* Positive test result at Screening for hepatitis B virus (defined as positive for hepatitis B surface antigen and/or hepatitis B core antibody).
* Previous exposure to BIIB074.
* Consumption of xanthine/caffeine-containing products (e.g., energy drinks, coffee, tea, caffeinated soda) within 48 hours of Day -1 and an unwillingness to refrain from product use during study participation.
* History of alcohol or substance abuse (as determined by the Investigator), a positive urine drug screen or alcohol breath test at Screening or Day -1, or an unwillingness to refrain from alcohol, or illicit or recreational drugs, during the study.
* History or evidence of habitual use of tobacco- or nicotine-containing products within 90 days of Screening, or a positive cotinine screen at Screening or Day -1.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PK of BIIB074 DCF to RCF as assessed by maximum observed concentration (Cmax) | Day 1, 2, 3, 8, 9, 10
PK of BIIB074 DCF to RCF as assessed by area under the concentration-time curve (AUC) from time 0 to time of the last measurable concentration (AUClast) | Day 1, 2, 3, 8, 9, 10
PK of BIIB074 DCF to RCF as assessed by AUC from time 0 to infinity (AUC∞) | Day 1, 2, 3, 8, 9, 10
PK of BIIB074 DCF as assessed by Cmax | Day 1, 2, 3, 8, 9, 10
PK of BIIB074 DCF as assessed by AUClast | Day 1, 2, 3, 8, 9, 10
PK of BIIB074 DCF as assessed by AUC∞ | Day 1, 2, 3, 8, 9, 10

SECONDARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 18
Number of participants with clinically significant laboratory assessment abnormalities | Up to Day 10
Number of participants with clinically significant vital sign abnormalities | Up to Day 10
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to Day 10
Number of participants with clinically significant physical examinations abnormalities | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Daytona Beach, Florida, United States